CLINICAL TRIAL: NCT05173155
Title: Comparison of Direct Anterior Approach vs. Lateral Hemiarthroplasty for Femoral Neck Fracture Repair: A Short-term Outcomes Study
Brief Title: Comparison of Direct Anterior Approach vs. Lateral Hemiarthroplasty for Femoral Neck Fracture Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210516-01H
Record Dates: First submitted 2021-11-09; First posted 2021-12-29 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patients will either receive a hemiarthroplasty in the direct anterior approach or the lateral approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct anterior approach for hemiarthroplasty (Experimental): Patients in this arm will receive a hemiarthroplasty using the direct anterior approach (DAA)
  Interventions: Procedure: surgical approach
- Lateral approach for hemiarthroplasty (Experimental): Patients in this arm will receive a hemiarthroplasty using the lateral approach
  Interventions: Procedure: surgical approach

INTERVENTIONS:
Procedure: surgical approach — Comparison of short-term outcomes (patient mobility, quality of life, function, pain, and safety parameters) for the direct anterior approach and Lateral approach for hemiarthroplasty for patients who have experienced a femoral-neck hip fracture.

SUMMARY:
Recent research has demonstrated that a hemiarthroplasty (replacement of half the joint) has lower rates of post-surgical complications than a total hip arthroplasty does. However, surgeons tend to vary in their approach to hemiarthroplasties. The lateral approach, which involves making an incision at the side of the patient's hip, requires surgeons to cut through the muscle to access the hip, which has been associated with greater muscle damage and slower rates of recovery. On the other hand, the direct anterior approach does not require the cutting of the patient's muscle and is therefore associated with minimal muscle damage and faster rates of recovery. This study will aim to assess the impact of the surgical approach (Direct Anterior Approach vs. Lateral approach) during hemiarthroplasty on patients' short-term mobility, quality of life, function, pain, and safety parameters.

DETAILED DESCRIPTION:
Hip fractures continue to increase with the aging Canadian population. Overall clinical and functional outcomes following hip fractures are poor, with only a third of patients returning to their pre-injury functional status (1). The hemiarthroplasty, which involves replacing the femoral head with a prosthesis after femoral neck fracture, is the procedure of choice in most intra-capsular hip fractures (2). Similar to the total hip arthroplasty, the hemiarthroplasty has been shown to be a safe and effective surgical technique. A recent study found that the hemiarthroplasty was associated with lower incidence of serious adverse events when compared to total hip arthroplasty (3). Approaches to the hip used by surgeons to perform arthroplasty procedures may vary. The lateral approach has been advocated by National bodies to be the approach of choice in arthroplasties for hip fractures because it is associated with a smaller dislocation compared to the posterior approach. However, the lateral approach is associated with significant morbidity to the musculature about the hip, which is already weak and degenerate in this population. Thus, the lateral approach may further impede recovery of this frail population. An attractive alternative of a surgical approach for this population may be the Direct Anterior Approach to the hip. This is an inter-nervous and inter-muscular approach, associated with minimal muscle damage. Furthermore, stability (i.e. dislocation risk) has been reported to be at least equal to that reported with the lateral approach. However, the Direct Anterior Approach is an approach associated with a learning curve of at least 100 cases and a potential increased risk of infection and peri-prosthetic fracture. The Direct Anterior Approach has shown to have superior outcomes compared to the lateral approach in total hip arthroplasty studies, however, no study to-date has compared these approaches in the setting of hip fractures where the lateral approach is considered the gold standard.

The investigators feel that this is an important question to answer and believe that The Ottawa Hospital has the appropriate expertise to conduct such study. This center has utilized the Direct Anterior Approach in total hip arthroplasty for the last 10 years and the team's extensive experienced has been published. At present, 5 arthroplasty surgeons routinely perform the Direct Anterior Approach for at least half of their hip arthroplasty patients. Furthermore, 3 of the staff surgeons are considered key opinion leaders on the Direct Anterior Approach having mentored many surgeons nationally and internationally in many teaching formats including courses and invited lectures.

The primary objective of this study is to assess the impact of the surgical approach for a hemiarthroplasty on patients' short-term mobility. The secondary objectives are to assess the impact of approach on quality of life, function, pain and safety parameters. The hypothesis is that the Direct Anterior Approach will lead to superior function and mobility at short-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a hemiarthroplasty for a femoral neck fracture;
* Patients capable of reading, writing and signing an informed consent form

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Short-term mobility | six days post-op
  The primary outcome measure will be mobility, assessed using the Short Physical Performance Battery (SPPB) test at post-operative day six or at discharge (4). This outcome assessed at this timeframe has been shown to be predictive of long-term function.

SECONDARY OUTCOMES:
EuroQol 5 | 2-weeks post-op
  Secondary outcomes measures will include evaluation of the patient's quality of life (using the EuroQol 5 questionnaire).
Visual Analogue Scale | 2-weeks post-op
  The Visual Analogue Scale will be given to patients 2- weeks post op to assess their levels of pain.
Opioid Use | 2-weeks post-op
  Opioid Use will be monitored for two weeks post-op via. phone calls and follow-up visits
Barthel 20 Index | ost-operative day six or at discharge, day 14, and week 6
  Family will be asked to complete questionnaires if patients are unable to. Activities of daily living (Barthel 20) will be assessed at post-operative day six or at discharge, day 14, and week 6 by a physiotherapist or nurse.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada